CLINICAL TRIAL: NCT03713762
Title: Anesthesia With Peribulbar Block: Lidocaine-bupivacaine vs Lidocaine-bupivacaine-fentanyl
Brief Title: Peribulbar Block: Lidocaine-bupivacaine vs Lidocaine-bupivacaine-fentanyl
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Medico Docente la Trinidad (Other)
Responsible Party: Principal Investigator, Leopoldo Wulff, Principal Investigator, anesthesiologist., Centro Medico Docente la Trinidad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBBCM
Record Dates: First submitted 2018-10-11; First posted 2018-10-22 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia, Local
Keywords: Peribulbar block
MeSH Terms: interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 LB (Experimental): Peribulbar block 1 was performed received 100 mg of lidocaine 5% and 15 mg of bupivacaine 0.5% for a total volume of the anesthetic mixture of 5 ml
  Interventions: Drug: peribulbar block 1 lidocaine/bupivacaine
- Group 2 LBF (Experimental): Peribulbar block 2 was performed received 100 mg of lidocaine 5%, 15 mg of 0.5% bupivacaine and 50 mcg of fentanyl citrate for a total volume of the anesthetic mixture of 6 ml.
  Interventions: Drug: peribulbar block 2 lidocaine/bupivacaine/fentanyl

INTERVENTIONS:
Drug: peribulbar block 1 lidocaine/bupivacaine — Peribulbar block: 100 mg of lidocaine 5% and 15 mg of bupivacaine 0.5% for a total volume of the anesthetic mixture of 5 ml.
  Other Names: lidocaine/bupivacaine
  Arms: Group 1 LB
Drug: peribulbar block 2 lidocaine/bupivacaine/fentanyl — Peribulbar block: 100 mg of lidocaine 5%, 15 mg of 0.5% bupivacaine and 50 mcg of fentanyl citrate for a total volume of the anesthetic mixture of 6 ml.
  Other Names: lidocaine/bupivacaine/fentanyl
  Arms: Group 2 LBF

SUMMARY:
Ophthalmological procedures such as cataract extraction can be carried out with a peribulbar block (PBB). The advantages of this anesthetic technique include a lower incidence of coughing, unwanted movements and emesis during awakening, in addition to providing adequate postoperative analgesia. The researchers want to investigate whether the use of fentanyl citrate by peribulbar route, when administered with a local anesthetic, shortens the anesthetic latency, interfere with the degree of akinesia and if provides greater postoperative analgesia.

DETAILED DESCRIPTION:
Article Type. Clinical trial study

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for cataract surgery (Cataract Extracapsular Extraction)
* With indication of regional anesthesia with peribulbar block
* Physical status ASA I or II
* Patients between 45 and 90 years of age

Exclusion Criteria:

* Allergic to amide-type anesthetics and fentanyl citrate
* Patients with a history of woody thorax
* Patients with uncompensated systemic diseases
* Patients in whom it was necessary to change the anesthetic technique due to insufficient analgesia or those in which the administration of intravenous analgesics was required during the operative period.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

PRIMARY OUTCOMES:
Latency period (lost of corneal reflex) | 10 minutes until the start of surgery
  lost of corneal reflex

SECONDARY OUTCOMES:
Ocular akinesia: movements of extraocular muscles | 10 minutes until the start of surgery
  movements of extraocular muscles
Incidence of postoperative pain | 2 Hours
  Analogous visual scale
postoperative complications | 2 hours
  bleeding or bruise

IPD SHARING:
Plan to Share IPD: Undecided